CLINICAL TRIAL: NCT02644954
Title: Assessing the Efficacy and Safety of Metformin in Treatment of Moderate Psoriasis: A Prospective Randomized Double Blind Controlled Study
Brief Title: Assessing the Efficacy and Safety of Metformin in Treatment of Moderate Psoriasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Sunil Dogra, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NK/1842/Res/1096
Record Dates: First submitted 2015-12-22; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Psoriasis
Keywords: psoriasis; Metformin
MeSH Terms: conditions — Psoriasis | interventions — Metformin; Coal Tar; calcipotriene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Active Comparator): Topical coal tar and topical calcipotriol + oral metformin 850mg twice daily
  Interventions: Drug: Metformin; Drug: Topical Coal tar; Drug: Topical calcipotriol
- Placebo (Placebo Comparator): Topical coal tar and topical calcipotriol
  Interventions: Drug: Placebo; Drug: Topical Coal tar; Drug: Topical calcipotriol

INTERVENTIONS:
Drug: Metformin — Metformin 850 mg twice daily given in the intervention arm to patients of moderate psoriasis
  Arms: Metformin
Drug: Placebo — Placebo drug twice daily given in the intervention arm to patients of moderate psoriasis
  Arms: Placebo
Drug: Topical Coal tar — Topical coal tar to be applied once daily
Drug: Topical calcipotriol — Topical calcipotriol to be applied once daily

SUMMARY:
Psoriasis vulgaris is a common, chronic, relapsing skin disease characterized by predominant involvement of skin, nails and joints. Recent advances in its patho-physiology have shifted the notion of psoriasis from that of a 'disease of the skin' to a 'T-cell mediated systemic disease'. Better understanding of its pathogenesis and co-morbidities along with the development of novel therapeutics like biological response modifiers has changed the way dermatologists approach the management of psoriasis. Based on the extent of involvement and effect on the quality of life, psoriasis may be mild to moderate in severity. This in turn forms the basis of treatment in majority of the patients. Topical therapies like coal tar, calcipotriol and corticosteroids are sufficient for mild and localized psoriasis. In more widespread or severe forms that are associated with significant decrease in quality of life of patient, phototherapy and systemic therapies are indicated either alone or in combination with each other. Although the introduction of biological therapies has revolutionized the treatment of psoriasis in recent years, such newer therapeutic options continue to elude the vast majority of patients in the developing and under developed world where the traditional agents like methotrexate, cyclosporine, acitretin and phototherapy still form the backbone of treatment.

The association of psoriasis with metabolic syndrome is now well documented. Metabolic syndrome is a cluster of risk factors including central obesity, atherogenic dyslipidemia, hypertension and glucose intolerance and is a strong predictor of cardiovascular diseases, diabetes and stroke. Metformin, an oral hypoglycemic agent of biguanide class is known for its multitude of action on various facets of metabolic syndrome. Recently it has also been found to inhibit keratinocyte proliferation in cell culture model of psoriasis.

The present study is designed as a randomized controlled double blind pilot study in which 40 patients with chronic plaque psoriasis of moderate severity (PASI ≥ 6 or DLQI ≥ 6) and metabolic syndrome (By modified ATP III criteria)4 or impaired glucose tolerance (defined as two-hour glucose levels of 140 to 199 mg per dL on the 75-g oral glucose tolerance test) will be recruited and randomized into two arms, A and B of 20 each, by using random number tables. Patients in arm A will be treated with topical anti-psoriatic treatment (including coal tar and vitamin D3 analogues only) and oral metformin 1g/day 850mg twice daily and patients in arm B will be treated with topical anti-psoriatic treatment and oral placebo tablets. Post randomization patients will be followed up at regular intervals for 24 weeks. During each visit, patients in both arms will be assessed for the severity of psoriasis by psoriasis activity severity index (PASI) and body mass index (BMI). Fasting blood glucose and insulin level, glycosylated haemoglobin (HbA1c) and parameters of metabolic syndrome (including waist circumference, fasting lipid profile and blood pressure) will be assessed at baseline and again at week 16 and 24. The primary aim of this study is to assess the efficacy and safety of oral metformin as an add on therapy for the treatment of chronic plaque psoriasis of moderate severity. The secondary aim is to assess the effect of metformin on parameters of the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Chronic plaque psoriasis of moderate severity, defined as PASI ≥ 6 and/or DLQI ≥ 6
* Metabolic syndrome (By modified ATP III criteria)4 or impaired glucose tolerance (defined as two-hour glucose levels of 140 to 199 mg per dL on the 75-g oral glucose tolerance test.)

Exclusion Criteria:

* Known drug allergies to biguanides.
* Psoriatic arthritis
* Pustular psoriasis
* Severe psoriasis PASI>10, DLQI> 10
* Patient with overt diabetes mellitus, defined as fasting blood sugar > 126mg/dl glucose tolerance test of >200mg/dl.
* Intake of oral hypoglycemic or systemic anti-psoriatic medication within the last 4 weeks.
* Patients on medications for cardiovascular, gastrointestinal, hepatic, renal, disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving 75% reduction in psoriasis activity severity index (PASI) | 1 year
  Evaluate the efficacy of oral metformin in chronic plaque psoriasis of moderate severity. The proportion of patients achieving PASI 75 assesses the efficacy.

SECONDARY OUTCOMES:
The proportion of patients achieving 90% reduction in psoriasis activity severity index (PASI) | 1 year
The number of patients who show change in parameters of metabolic syndrome after taking metformin | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Dogra, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh

REFERENCES:
- [Background] Torti DC, Feldman SR. Interleukin-12, interleukin-23, and psoriasis: current prospects. J Am Acad Dermatol. 2007 Dec;57(6):1059-68. doi: 10.1016/j.jaad.2007.07.016. Epub 2007 Aug 15. PMID 17706835
- [Background] Li W, Ma W, Zhong H, Liu W, Sun Q. Metformin inhibits proliferation of human keratinocytes through a mechanism associated with activation of the MAPK signaling pathway. Exp Ther Med. 2014 Feb;7(2):389-392. doi: 10.3892/etm.2013.1416. Epub 2013 Nov 19. PMID 24396411
- [Background] Reich K. The concept of psoriasis as a systemic inflammation: implications for disease management. J Eur Acad Dermatol Venereol. 2012 Mar;26 Suppl 2:3-11. doi: 10.1111/j.1468-3083.2011.04410.x. PMID 22356630
- [Background] Spah F. Inflammation in atherosclerosis and psoriasis: common pathogenic mechanisms and the potential for an integrated treatment approach. Br J Dermatol. 2008 Aug;159 Suppl 2:10-7. doi: 10.1111/j.1365-2133.2008.08780.x. PMID 18700910
- [Background] Gisondi P, Tessari G, Conti A, Piaserico S, Schianchi S, Peserico A, Giannetti A, Girolomoni G. Prevalence of metabolic syndrome in patients with psoriasis: a hospital-based case-control study. Br J Dermatol. 2007 Jul;157(1):68-73. doi: 10.1111/j.1365-2133.2007.07986.x. Epub 2007 Jun 6. PMID 17553036
- [Background] Gelfand JM, Neimann AL, Shin DB, Wang X, Margolis DJ, Troxel AB. Risk of myocardial infarction in patients with psoriasis. JAMA. 2006 Oct 11;296(14):1735-41. doi: 10.1001/jama.296.14.1735. PMID 17032986
- [Background] Ludwig RJ, Herzog C, Rostock A, Ochsendorf FR, Zollner TM, Thaci D, Kaufmann R, Vogl TJ, Boehncke WH. Psoriasis: a possible risk factor for development of coronary artery calcification. Br J Dermatol. 2007 Feb;156(2):271-6. doi: 10.1111/j.1365-2133.2006.07562.x. PMID 17223866
- [Background] Ouchi N, Kihara S, Arita Y, Maeda K, Kuriyama H, Okamoto Y, Hotta K, Nishida M, Takahashi M, Nakamura T, Yamashita S, Funahashi T, Matsuzawa Y. Novel modulator for endothelial adhesion molecules: adipocyte-derived plasma protein adiponectin. Circulation. 1999 Dec 21-28;100(25):2473-6. doi: 10.1161/01.cir.100.25.2473. PMID 10604883
- [Background] Pathirana D, Ormerod AD, Saiag P, Smith C, Spuls PI, Nast A, Barker J, Bos JD, Burmester GR, Chimenti S, Dubertret L, Eberlein B, Erdmann R, Ferguson J, Girolomoni G, Gisondi P, Giunta A, Griffiths C, Honigsmann H, Hussain M, Jobling R, Karvonen SL, Kemeny L, Kopp I, Leonardi C, Maccarone M, Menter A, Mrowietz U, Naldi L, Nijsten T, Ortonne JP, Orzechowski HD, Rantanen T, Reich K, Reytan N, Richards H, Thio HB, van de Kerkhof P, Rzany B. European S3-guidelines on the systemic treatment of psoriasis vulgaris. J Eur Acad Dermatol Venereol. 2009 Oct;23 Suppl 2:1-70. doi: 10.1111/j.1468-3083.2009.03389.x. PMID 19712190
- [Background] Solomon DH, Massarotti E, Garg R, Liu J, Canning C, Schneeweiss S. Association between disease-modifying antirheumatic drugs and diabetes risk in patients with rheumatoid arthritis and psoriasis. JAMA. 2011 Jun 22;305(24):2525-31. doi: 10.1001/jama.2011.878. PMID 21693740
- [Background] Jensterle M, Janez A, Mlinar B, Marc J, Prezelj J, Pfeifer M. Impact of metformin and rosiglitazone treatment on glucose transporter 4 mRNA expression in women with polycystic ovary syndrome. Eur J Endocrinol. 2008 Jun;158(6):793-801. doi: 10.1530/EJE-07-0857. Epub 2008 Mar 5. PMID 18322300
- [Background] Mourao-Junior CA, Sa JR, Guedes OM, Dib SA. Effects of metformin on the glycemic control, lipid profile, and arterial blood pressure of type 2 diabetic patients with metabolic syndrome already on insulin. Braz J Med Biol Res. 2006 Apr;39(4):489-94. doi: 10.1590/s0100-879x2006000400009. Epub 2006 Apr 3. PMID 16612472
- [Background] Viollet B, Guigas B, Sanz Garcia N, Leclerc J, Foretz M, Andreelli F. Cellular and molecular mechanisms of metformin: an overview. Clin Sci (Lond). 2012 Mar;122(6):253-70. doi: 10.1042/CS20110386. PMID 22117616
- [Background] Hadi NR, Al-Amran FG, Swadi A. Metformin ameliorates methotrexate-induced hepatotoxicity. J Pharmacol Pharmacother. 2012 Jul;3(3):248-53. doi: 10.4103/0976-500X.99426. PMID 23129960
- [Background] Charles MA, Morange P, Eschwege E, Andre P, Vague P, Juhan-Vague I. Effect of weight change and metformin on fibrinolysis and the von Willebrand factor in obese nondiabetic subjects: the BIGPRO1 Study. Biguanides and the Prevention of the Risk of Obesity. Diabetes Care. 1998 Nov;21(11):1967-72. doi: 10.2337/diacare.21.11.1967. PMID 9802752
- [Background] Batchuluun B, Inoguchi T, Sonoda N, Sasaki S, Inoue T, Fujimura Y, Miura D, Takayanagi R. Metformin and liraglutide ameliorate high glucose-induced oxidative stress via inhibition of PKC-NAD(P)H oxidase pathway in human aortic endothelial cells. Atherosclerosis. 2014 Jan;232(1):156-64. doi: 10.1016/j.atherosclerosis.2013.10.025. Epub 2013 Nov 5. PMID 24401231
- [Background] Glossmann H, Reider N. A marriage of two "Methusalem" drugs for the treatment of psoriasis?: Arguments for a pilot trial with metformin as add-on for methotrexate. Dermatoendocrinol. 2013 Apr 1;5(2):252-63. doi: 10.4161/derm.23874. PMID 24194965